CLINICAL TRIAL: NCT03507049
Title: Sacroiliac Joint Fusion Versus Sham Operation for Treatment of Sacroiliac Joint Pain. A Prosepctive Double Blinded Randomized Controlled Multicenter Trial.
Brief Title: Sacroiliac Joint Fusion Versus Sham Operation for Treatment of Sacroiliac Joint Pain
Acronym: SIFSO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Johan Kibsgård, Senior consultant, associated professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/1892 A
Record Dates: First submitted 2018-04-06; First posted 2018-04-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Sacroiliac Joint Somatic Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing sacroiliac joint fusion and sham surgery. A prospective double blinded randomized controlled multicenter trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Active Comparator): The intervention Group receives operation with SI-joint arthrodesis with the iFuse implant. The patient undergoes full anesthesia. The procedure starts with an approximately 5cm long skin incision over the posterolateral aspect of the pelvis. A guide-pin is inserted over the sacroiliac joint at the desired entry-point, verified by fluoroscopy. The surgeons drills and boraches over the pin and the ifuse implant is inserted. This is repeated for a total of three implants. The wound is closed with non-resorbable suture. An injection of the SIJ with local anesthetic is performed under guidance of fluoroscopy at the time of the procedure.
  Interventions: Procedure: iFuse
- Sham group (Sham Comparator): The sham operation will consist of the surgeon making the same skin incision as for an iFuse procedure, although nothing more, and then closing the wound.
  The patients undergoing a sham operation will be under general anesthesia for a random time of 20-40minutes in order to keep the two procedures as similar as possible.
  An injection of the SIJ with local anesthetic is performed under guidance of fluoroscopy at the time of the procedure.
  Interventions: Procedure: sham group
- Functional MRI study (Other): The Swedish patients will also undergo quantitative sensory testing at inclusion and at 6 month follow-up. At the same time they will undergo a cerebral MRI and a Functional MRI looking at activation of the CNS from pain in the sacroiliac joints induced by one leg lift. The purpose of this study is to look at contributing factors in treatment response. One hopes to map which CNS mechanisms are involved in causing the chronic pain these patients experience as well as how they respond to treatment.
  Interventions: Radiation: fMRI study

INTERVENTIONS:
Procedure: iFuse — ifuse will be implanted as described in section on the active comparator arm of the study.
  Other Names: SI Bone iFuse
  Arms: Intervention group
Procedure: sham group — sham surgery will be performed as desrcribed in section on sham comparator.
  Other Names: Sham surgery
  Arms: Sham group
Radiation: fMRI study — Quantitative sensory testing, cerebral MRI and functional MRI will be done to examine pain mechanism and activation in the central nervous system.
  Arms: Functional MRI study

SUMMARY:
Sacroiliac joint fusion versus sham operasjon for treatment of sacroiliac pain. A prospective double blinded randomized controlled multicentre study.

DETAILED DESCRIPTION:
Sacroiliac(SI) joint pain can lead to long-lasting severe pain and reduce physical function. It is shown to be the source of pain in 13-30% of patients with low back pain. Former surgical techniques had a high level of complications and low success rates. Newer mini-invasive surgical approaches have shown promising results in scientific studies. It is difficult to find an adequate control group for surgery as most patients already have tried conservative and alternative treatments without effect. A sham-designed study is the best alternative. This study is designed as a prospective randomized double blinded controlled mulitcenter trial. The investigators want to examine whether there is a difference in SI joint pain in patients operated with miniinvasive arthrodesis of the SI joint compared to a sham operated control group. Patients with SI joint pain are included. They will be randomized to either surgery with arthrodesis or sham surgery. Neither patient nor health personell who work with the patient after the surgery will know what has been done. The primary end point for the study is group difference in sacroiliac joint pain on the operated side after 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 at time of screening
2. Patient with suspected SIJ pain for >6 months or >18 months for pregnancy induced pelvic girdle pain.
3. Diagnosis of the SI joint as the primary pain generator based on ALL of the following:

A. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test)

B. Patient has at least 3 of 6 physical examination maneuvers specific for SI joint pain:

1. Compression
2. Posterior Pelvic Pain Provocation test - P4 (Thigh Thrust)
3. Palpation of the long dorsal ligament
4. Patrick's test (Faber)
5. Leg Raise (ASLR )
6. Geanslens test

C. Patient has improvement in lower back pain NRS of at least 50% of the pre injection NRS score after fluoroscopic controlled injection of local anesthetic into affected SI joint (including previous documented test <6 months ago)

4. Baseline Oswestry Disability Index (ODI) score of at least 30%

5. Baseline lower back pain score of at least 5 on 0-10 point NRS

6. Patient should have tried adequate forms of conservative treatment with little or no response.

7. Patient has signed study-specific informed consent

8. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements.

9. Patients with unilateral or bilateral pain can be included in the study if they clearly can differentiate between the two sides. It is the most painful side that will be included and randomized to SIJ fusion or sham surgery in the study.

Exclusion Criteria:

1. Severe low back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture.
2. Sacroiliac pathology caused by auto-immune disease (e.g. ankylosing spondylitis) and/or neoplasia (e.g. benign or malignant tumor) and/or crystal arthropathy
3. History of recent (<1 year) fracture of the pelvis with documented malunion, non-union of sacrum or ilium or any type of internal fixation of the pelvic ring.
4. Spine surgery during the past 12 months.
5. Previously diagnosed or suspected osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture)
6. Documented osteomalacia or other metabolic bone disease
7. Any condition or anatomy that makes treatment with the iFuse Implant System infeasible
8. Patients with prior successful fusion to the contra lateral side are exluded from the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2030-05-25 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure - Numeric Rating Scale operated side | 6 months
  the primary endpoint is group difference in Numeric Rating Scale(NRS) pain-score on the operated side at six months postoperatively. Numeric rating scale is a pain-score scale from 0-10, where 0 is no pain and 10 is worst possible pain.

SECONDARY OUTCOMES:
Baseline NRS | baseline, 3, 6, 12 and 24 months
  Change from baseline Numeric Rating Scale (NRS) pain-score on the operated side at 3,6,12 and 24 months
Global NRS | baseline,3 ,6 ,12 ,24 months
  Change from baseline global NRS at 3,6,12 and 24 months
NRS on non-operated side | baseline, 3, 6, 12, 24 months
  Change from baseline in non-operated side NRS at 3,6,12 and 24 months
NRS leg pain | baseline, 3,6,12,24 months
  Change from baseline leg pain NRS at 3,6,12,24 months
Oswestry disability index (ODI) | baseline, 3, 6,12, 24 months
  Change in disability due to pelvic pain measured by Oswestry Disability Index(ODI) at 3,6,12,24 months
Pelvic girdle questionnaire | baseline, 3, 6, 12, 24 months
  Change in disability due to pelvic pain measured by Pelvic Girdle Questionnaire(PGQ) at 3,6,12,24 months
Quality of life (EQ-5D) | baseline, 3, 6, 12, 24 months
  Change in quality of life measured by EQ-5D at 3,6,12,24 months
Device breakage, loosening or migration on CT of the sacroiliac joint | 12 months
  Device breakage loosening or migration at 12 months judged by clinical symptoms and CT of the sacroiliac joint.

OTHER OUTCOMES:
Adverse events | 3,6,12,24 months
  registration of any adverse events after procedure completed
Change in Compression test of the sacroiliac joint | baseline, 3, 6,12, 24 months
  Change in compression test of the sacroiliac joint which is an objective clinical test. Outcome is negative or positive test dependent on whether pain is provoked or not in the sacroiliac joint.
Change in Posterior Pelvic Pain Provocation (P4) test of the sacroiliac joint | baseline, 3, 6,12, 24 months
  Change in Posterior Pelvic pain Provocation (P4) test of the sacroiliac joint which is an objective clinical test. Outcome is negative or positive test dependent on whether pain is provoked or not in the sacroiliac joint.
Change in Palpation of long dorsal ligament as test of the sacroiliac joint | baseline, 3, 6,12, 24 months
  Change in Palpation of long dorsal ligament as test of the sacroiliac joint which is an objective clinical test. Outcome is negative or positive test dependent on whether pain is provoked or not along the ligament.
Change in Patricks (FABER) test of the sacroiliac joint | baseline, 3, 6,12, 24 months
  Change in Patricks (FABER) test of the sacroiliac joint which is an objective clinical test. Outcome is negative or positive test dependent on whether pain is provoked or not in the sacroiliac joint. .
Change in active straight leg raise test (ASLR) of the sacroiliac joint | baseline, 3, 6,12, 24 months
  Change in active straight leg raise test(ASLR) of the sacroiliac joint which is an objective clinical test. Results are recorded on a grad 0 to 5, where not difficult at all = 0; minimally difficult = 1; somewhat difficult = 2; fairly difficult = 3; very difficult = 4; unable to do = 5.
Change in Gaenslens test | baseline, 3, 6,12, 24 months
  Change in Gaenslens test which is an objective clinical tests for the sacroiliac joint. Outcome is recorded as positive or negative test dependent on whether pain is provoked or not in the sacroiliac joint.
6 minute walk test to record ambulatory status | baseline, 3, 6,12, 24 months.
  Patients will be tested with 6minute walk test to test ambulatory status. The test is performed by marking a distance equal to 50meters. The patient is instructed to walk back and forth between the marks as quickly and as many times as they manage in 6 minutes. The total distance walked is recorded.
Timed up and og test to record ambulatory status | baseline, 3, 6,12, 24 months.
  Patients will be tested with Timed up and go, to test ambulatory status.Timed up and go test the time it takes the patient to get up from a Chair, walk 3 meters and back and be seated again.
Work status | baseline, 3, 6,12, 24 months.
  Patients will be asked to fill out standardized questionnaire on work status

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Johan Dr Kibsgård, PhD, MD, Principal Investigator — Oslo University Hospital; Paul Dr Gerdhem, PhD, MD, Study Chair — Karolinska University Hospital
Locations (2):
- Rikshospitalet, Oslo University Hospital, Oslo, Norway
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Randers EM, Gerdhem P, Stuge B, Diarbakerli E, Nordsletten L, Rohrl SM, Kibsgard TJ. The effect of minimally invasive sacroiliac joint fusion compared to sham operation: a double-blind randomized placebo-controlled trial. EClinicalMedicine. 2024 Feb 1;68:102438. doi: 10.1016/j.eclinm.2024.102438. eCollection 2024 Feb. PMID 38328752

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03507049/Prot_SAP_000.pdf